CLINICAL TRIAL: NCT00666354
Title: Phase IIB Dose Response and Safety Study of Topical Formulations of Methotrexate (MQX-5902, MQX-5904 and MQX-5906) in the Treatment of Fingernail Psoriasis
Brief Title: Dose Response and Safety Study of Topical Methotrexate for the Treatment of Fingernail Psoriasis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: MediQuest Therapeutics (Industry)
Responsible Party: Fred Dechow/President and CEO, MediQuest Therapeutics
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06-003; ISRCTN62739763
Record Dates: First submitted 2008-04-22; First posted 2008-04-24 (Estimated); Last update posted 2009-02-10 (Estimated); Status verified 2009-02

CONDITIONS: Fingernail Psoriasis
Keywords: Nail Psoriasis; Psoriasis; Fingernail Psoriasis; Methotrexate
MeSH Terms: conditions — Psoriasis | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator)
  Interventions: Drug: Methotrexate
- 2 (Active Comparator)
  Interventions: Drug: Methotrexate
- 3 (Active Comparator)
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Methotrexate — 0.01 gram of topical amphimatrix containing 0.05% methotrexate per affected nail and adjacent skin folds applied daily for three months.
  Other Names: MQX-5906
  Arms: 1
Drug: Methotrexate — 0.01 gram of topical amphimatrix containing 0.25% methotrexate per affected nail and adjacent skin folds applied daily for three months.
  Other Names: MQX-5902
  Arms: 2
Drug: Methotrexate — 0.01 gram of topical amphimatrix containing 1.0% methotrexate per affected nail and adjacent skin folds applied daily for three months.
  Other Names: MQX-5904
  Arms: 3

SUMMARY:
The purpose of this clinical study is to compare the efficacy and safety of three concentrations of topical methotrexate for the treatment of fingernail psoriasis.

DETAILED DESCRIPTION:
The purpose of this clinical study is to compare, in a controlled fashion, the response to three concentrations of methotrexate in novel topical formulations in the treatment of subjects with psoriasis of the fingernails. Such a determination will be used as the basis for evidence of efficacy and safety of these formulations as a therapeutic treatment for fingernail psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed moderate fingernail psoriasis of at least two fingernails.
* Stable and unchanged psoriasis therapies for 2 months and must not have received methotrexate for 3 months prior to screening.
* Female patients who are not 5 years post menopausal or surgically sterile must use appropriate birth control for specified time periods and have negative pregnancy tests.

Exclusion Criteria:

* Target or control fingernails that are thicker than 2mm, abnormal or infected (bacterial or fungal).
* Patients with immunosuppression, HIV, or neuropathies of the hand.
* Use of any methotrexate preparation, any topical anti-psoriatic medications or ultraviolet treatment within 2 months of study visit 1.
* Use of more that one 2-week course of oral corticosteroid therapy or one injection during 3 months prior to the screening visit.
* Use of manicures or cosmetic nail products during and within 7 days of the start of treatment.
* Use of any drug known to have potential for toxicity to a major organ during and within 90 days prior to the start of treatment.
* Patients who are nursing, pregnant or plan to become pregnant or father a child within the study time frame including within three months of the last dose of study medication.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2007-10; Primary Completion 2008-09 (Estimated); Study Completion 2009-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate improvements in the appearance of the target fingernail, utilizing photography for imaging and independent photograph evaluators. | Monthly

SECONDARY OUTCOMES:
Improvement in appearance of the control fingernail, improvement of the target fingernail using mNAPSI (a modification of the Nail Psoriasis Severity Index), and comparison of improvement of mNAPSI of the target and control fingernails. | Monthly
Information on the relative changes in nail psoriasis severity of the other affected fingernails will be collected. | Monthly
Comparison of nail growth of the target and control fingernails as determined from nail notch movement measured on nail photographs will be performed. | Monthly
Assess safety, i.e., the frequency and severity of adverse events associated with MQX-5902, MQX-5904 and MQX-5906 in the treatment of patients with fingernail psoriasis. | Monthly

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Neil McHugh, Principal Investigator — Royal National Hospital for Rheumatic Diseases
Locations (7):
- United Kingdom (7):
  - University of Manchester, The Dermatology Centre, Salford, Manchester
  - Great Western Hospital Rheumatology Department, Swindon, Wiltshire
  - Aberdeen Royal Infirmary Dermatology Outpatients Clinic, Aberdeen
  - Royal National Hospital for Rheumatic Diseases, Bath
  - University Hospital of Wales, Welsh Institute of Dermatology, Cardiff
  - Leeds General Infirmary Department of Dermatology, Leeds
  - George Eliot Hospital, Department of Dermatology, Nuneaton